CLINICAL TRIAL: NCT06855823
Title: A Phase I/II, Open-Label Clinical Trial to Evaluate the Efficacy and Safety of Golidocitinib As Monotherapy or in Combination with Pomalidomide for the Treatment of Relapsed/Refractory Peripheral T-Cell Lymphoma (R/R PTCL)
Brief Title: A Phase I/II Study of Golidocitinib Combined with Pomalidomide in R/R PTCL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2024-807-01
Record Dates: First submitted 2025-01-16; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory Peripheral T-Cell Lymphoma (R/R PTCL)
Keywords: Golidocitinib; Pomalidomide; Relapsed/Refractory PTCL
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Golicitinib combined with Pomadomide in the treatment of R/R PTCL (Experimental): Combination therapy: Subjects received Golidocitinib 150 mg orally once daily continuously, plus Pomalidomide at three dose levels (2 mg, 3 mg, 4 mg) orally on days 1-21 of each 28-day cycle. The dose of Pomalidomide will be escalated according to the 3+3 design to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D). The treatment will continue until disease progression, intolerable toxicity, withdrawal of consent, or other criteria for discontinuation are met, with a maximum treatment duration of 2 years.
  Interventions: Drug: Golicitinib combined with Pomadomide

INTERVENTIONS:
Drug: Golicitinib combined with Pomadomide — golidoctinib 150 mgqd, pomalidomide 2mg/3mg/4mgqd
  Other Names: Golidocitinib: JAK1 Inhibitor; Pomalidomide: Third-generation Immunomodulatory Drug (IMiD)

SUMMARY:
This is a phase I/II clinical trial to evaluate the efficacy and safety of Golidocitinib combined with Pomalidomide for relapsed/refractory peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
This clinical trial aims to investigate the efficacy and safety of Golidocitinib combined with Pomalidomide in treating relapsed/refractory peripheral T-cell lymphoma (R/R PTCL). The study is a prospective, open-label, phase I/II clinical trial initiated by investigators. It plans to enroll approximately 26-33 patients who have not previously received Golidocitinib or Pomalidomide. The primary endpoint for phase I is to assess the dose-limiting toxicity (DLT) of Pomalidomide in combination with Golidocitinib, estimate the maximum tolerated dose (MTD), and determine the recommended phase II dose (RP2D). For phase II, the primary endpoint is to evaluate the objective response rate (ORR) of the combination therapy. Secondary endpoints include duration of response (DOR), complete response rate (CR), progression-free survival (PFS), overall survival (OS), time to response (TTR), and safety indicators. The study will provide valuable data on the potential benefits and risks of this novel combination therapy for R/R PTCL patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must demonstrate a comprehensive understanding of the study protocol, voluntarily consent to participation, and execute the informed consent document.
* Inclusive of both genders, participants must be aged 18 years or older and not exceed 80 years of age.
* Histopathological confirmation of peripheral T-cell lymphoma (PTCL) must adhere to the World Health Organization (WHO) 2016 classification criteria. This encompasses a range of PTCL subtypes, including but not limited to peripheral T cell lymphoma not otherwise specified (PTCL NOS), vascular immunoblastic T cell lymphoma (AITL), NK/T cell lymphoma, anaplastic large cell lymphoma ALK positive (ALCL ALK+), anaplastic large cell lymphoma ALK negative (ALCL ALK-), enteropathy-associated T-cell lymphoma, hepato-splenic T-cell lymphoma, subcutaneous panniculitis-like T-cell lymphoma, and other subtypes deemed eligible for study participation by the investigators.
* Subjects must exhibit relapsed or refractory disease following prior systemic therapy, which may include autologous hematopoietic stem cell transplantation. Relapse is characterized by disease recurrence post-complete response (CR), whereas refractory disease is indicated by stable disease (SD) or progressive disease (PD) following systemic chemotherapy, or by the absence of CR upon treatment completion necessitating further intervention.
* At least one lesion must be present that is evaluable or measurable according to the Lugano2014 criteria: for lymph node lesions, the minimum measurable length is 1.5cm; for non-lymph node lesions, extra-nodal lesions must exceed 1.0cm in length.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status score ranging from 0 to 2.
* Laboratory parameters must meet the following criteria: (1) absolute neutrophil count (ANC) of at least 1.5×10^9/L; (2) platelet count (PLT) of at least 75×10^9/L (with a minimum of 50×10^9/L for patients with bone marrow infiltration); (3) hemoglobin (HB) level of at least 80 g/L; (4) serum total bilirubin (TBIL) not exceeding 1.5 times the upper limit of normal (ULN); (5) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels not exceeding 2.5 times the ULN; (6) serum creatinine (Scr) not exceeding 1.5 times the ULN.
* Participants must not have undergone radiotherapy, chemotherapy, targeted therapy, or hematopoietic stem cell transplantation within the 3 weeks preceding study enrollment.
* Investigators must assess that the subject has a life expectancy of at least six months.

Exclusion Criteria:

* Presence of hemophagocytic syndrome.
* Involvement of the central nervous system or meninges by lymphoma.
* A history of malignant tumors within the past five years, with the exception of locally curable tumors that have been subjected to radical treatment (e.g., basal or squamous cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast).
* History of any of the following treatments:(1) Allogeneic hematopoietic stem cell transplantation prior to the administration of the investigational drug; (2) Autologous hematopoietic stem cell transplantation within six months preceding study drug administration; (3) Previous use of golidocitinib or pomalidomide; (4) Current use of vitamin K antagonists, antiplatelet drugs, anticoagulants (or unable to discontinue within one week prior to study commencement); (5) Requirement for systemic glucocorticoid therapy or other immunosuppressive therapy for any condition within 14 days prior to study initiation; topical, ocular, intraarticular, intranasal, and inhaled glucocorticoids are permitted; short-term (≤7 days) glucocorticoid use for prophylactic treatment or non-autoimmune diseases is allowed; (6) Cytotoxic chemotherapy must not have been terminated within 21 days before the start of the study; (7) Received systemic antineoplastic therapy (including macromolecular monoclonal antibodies and immunotherapy drugs) within four weeks of study initiation; (8) Undergone major surgery (excluding vascular access surgery) or experienced serious trauma within four weeks before the start of the study; or received radiation therapy within three weeks; (9) Received other toxin/isotope-immune antibody conjugates within ten weeks; (10) For other types of new drug use, the researcher shall make a determination after comprehensive assessment; (11) Received an experimental drug or investigational drug in another trial within 30 days prior to study commencement; (12) Received live vaccines (except attenuated influenza vaccines) 28 days prior to study drug administration.
* Active infections, including: (1) Known active/latent tuberculosis, including a positive tuberculin skin test or findings on plain chest X-ray/CT (positive skin test results should exhibit an induration diameter greater than 10 mm, or as per local clinical criteria); (2) Known history of Human Immunodeficiency Virus (HIV) infection and/or acquired immunodeficiency syndrome; (3) Patients with active chronic hepatitis B or hepatitis C. Hepatitis B Surface Antigen (HBsAg) must be further tested with Hepatitis B Virus (HBV) DNA titer (not to exceed 1000 IU/mL) at the screening stage. Enrollment in the trial is only possible after excluding active hepatitis B or C infections requiring treatment. Hepatitis B carriers, patients with stable hepatitis B after drug treatment (with a DNA titer not exceeding 1000 IU/mL), and cured hepatitis C patients are eligible for enrollment. (For included hepatitis B patients, entecavir and other anti-hepatitis B virus treatments should be administered orally as per guidelines); (4) Active viral infections other than hepatitis B and C (e.g., herpes zoster, cytomegalovirus); (5) Infections necessitating oral or intravenous antimicrobial therapy; (6) Bacterial infections within 30 days, including pneumonia.
* Active autoimmune diseases requiring systemic treatment within the past two years (hormone replacement therapy not considered systemic treatment, such as type I diabetes, hypothyroidism managed with thyroxine replacement alone, adrenal or pituitary insufficiency requiring only physiological glucocorticoid replacement); patients with autoimmune diseases not requiring systemic treatment in the past two years may be enrolled.
* Uncontrolled cardiac clinical symptoms or diseases, such as: i. New York Heart Association (NYHA) class > 2 heart failure ii. Unstable angina pectoris iii. Myocardial infarction within one year iv. Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* Prior interstitial lung disease (except for asymptomatic interstitial lung disease induced by radiotherapy).
* Presence of unresolved adverse drug reactions greater than CTCAE grade 1 (excluding alopecia) before study initiation.
* Patients with hypersensitivity to golidocitinib or pomalidomide/capsule excipients or other chemical analogs; patients with a known history of severe allergic reactions to monoclonal antibodies (CTCAE≥3) and uncontrolled allergic asthma.
* Subjects requiring supportive treatment for refractory nausea, vomiting, chronic gastrointestinal disorders, dysphagia, or prior surgical removal of intestinal segments that may impede adequate drug absorption.
* Pregnant and lactating women and individuals of childbearing age who are unwilling to practice contraceptive measures.
* Individuals with psychiatric illnesses or those incapable of providing informed consent.
* Deemed ineligible for study participation by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD) in Phase I | Up to approximately 1 month
  Incidence of dose-limiting toxicities during the first cycle of treatment and determination of the maximum tolerated dose of pomalidomide in combination with golidocitinib.
Objective Response Rate (ORR) in Phase II | Up to approximately 24 months
  The proportion of patients achieving either complete response (CR) or partial response (PR) as per the 2014 Lugano criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) after 4 cycles (Lugano 2014) | Up to approximately 2 years
  ORR is defined as the proportion of subjects achieving complete response (CR) or partial response (PR).
Complete Response Rate (CRR) after 4 cycles (Lugano 2014) | Up to approximately 2 years
  CRR is calculated as the percentage of the sum of the number of patients in complete remission (CR) and complete remission without confirmation (CRu) to the total number of patients in the full analysis set.
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first documentation of confirmed response (CR or PR) to the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the first dose of investigational products until documentation of PD or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from the first dose of investigational products until death due to any cause.
Incidence and Severity of Adverse Events (AEs) | Up to approximately 2 years
  The incidence and severity of AEs are assessed to evaluate the safety profile of golidocitinib combined with pomalidomide.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China